CLINICAL TRIAL: NCT00096109
Title: A Phase II Clinical Trial of 17-Allyamino-17-Demethoxygeldanamycin (17-AAG) in Chemotherapy Refractory Metastatic Breast Cancer
Brief Title: Tanespimycin in Treating Women With Refractory Locally Advanced or Metastatic Breast Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Closed to accrual before all 12 planned patients were enrolled.
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-03058; C-2803; U01CA062502 (NIH); U01CA062487 (NIH); CDR0000391198 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 2004-11-09; First posted 2004-11-09 (Estimated); Results first posted 2017-01-16 (Estimated); Last update posted 2017-01-16 (Estimated); Status verified 2016-11

CONDITIONS: Recurrent Breast Cancer; Stage IIIB Breast Cancer; Stage IIIC Breast Cancer; Stage IV Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — tanespimycin

ARMS (1):
- Treatment (tanespimycin) (Experimental): Patients receive tanespimycin IV over 1-6 hours on days 1, 4, 8, and 11. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: tanespimycin; Other: laboratory biomarker analysis

INTERVENTIONS:
Drug: tanespimycin — Given IV
  Other Names: 17-AAG
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
This phase II trial is studying how well tanespimycin works in treating women with refractory locally advanced or metastatic breast cancer. Drugs used in chemotherapy, such as tanespimycin, work in different ways to stop tumor cells from dividing so they stop growing or die

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the response rate of 17-Allylamino-17-Demethoxygeldanamycin (17-AAG) (tanespimycin) in patients with refractory/resistant metastatic breast cancer.

II. To determine the progression free survival (PFS) of patients with refractory/resistant metastatic breast cancer when treated with 17-AAG.

III. To correlate patients' her2/neu status with response to 17-AAG treatment.

OUTLINE: This is a multicenter study.

Patients receive tanespimycin IV over 1-6 hours on days 1, 4, 8, and 11. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.

Patients are followed at day 30, every 10-12 weeks until disease progression, and then every 3 months thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Primary adenocarcinoma of the breast confirmed by histology or cytology
* Locally advanced or metastatic disease not amenable to surgery or radiation therapy with curative intent
* At least 1 measurable (target) lesion (i.e. any malignant tumor mass that can be accurately measured in at least 1 dimension of >= 2 cm with conventional radiographic techniques or >= 1 cm with magnetic resonance imaging [MRI] or spiral computerized tomography [CT] scans), not previously irradiated
* Progressive disease following hormonal therapy in appropriate patients (ER-positive and/or indolent disease)
* Progressive disease following treatment with both an anthracycline and a taxane (as adjuvant therapy or for metastatic disease) or contraindication to such treatment
* All previous cytotoxic chemotherapy must have been discontinued at least 4 weeks before study entry and all acute toxicity of prior therapy (excluding alopecia and neurotoxicity) must be resolved to NCI CTC (Version 3.0) grade =< 1; patients must have discontinued treatment with nitrosoureas or mitomycin C at least 6 weeks prior to study entry
* All previous hormonal therapy must have been discontinued for at least 2 weeks before study entry
* Life expectancy of >= 3 months
* ECOG performance status (PS) of 0-2
* Absolute neutrophil count (ANC) >= 1500/mm^3
* Platelets >= 100,000/mm^3
* Hemoglobin >= 9.0 g/dL
* Creatinine (Cr) =< upper limit of normal (ULN) or Cr Clearance > 60 mL/min/m^2
* Total bilirubin =< 1.5X ULN
* Alanine aminotransferase (ALT) =< 1.5X ULN or =< 3X ULN with liver metastases
* Aspartate aminotransferase (AST) =< 5X ULN or =< 3X ULN with liver metastases
* Negative serum pregnancy test within 7 days of enrollment for pre-menopausal women or women within 6 months of menopause
* Willingness and ability to comply with scheduled visits, treatment plan, laboratory tests, and other study procedures
* Evidence of a personally signed and dated informed consent document indicating that the patient (or a legally acceptable representative) has been informed and understands all pertinent aspects and the investigational nature of the trial

Exclusion Criteria:

* Current treatment with any other anti-neoplastic agent, including trastuzumab; patients may continue to receive zoledronic acid for bone metastases or hypercalcemia
* Radiation therapy within 2 weeks of enrollment or surgery within 4 weeks
* Known brain or leptomeningeal metastatic disease requiring active therapy; (Patients with asymptomatic previously treated metastases to these areas are eligible)
* Any of the following conditions within 6 months of enrollment: myocardial infarction, severe/unstable angina, symptomatic congestive heart failure, cerebrovascular accident or transient ischemic attack, coronary/peripheral artery bypass grafting; patients who have experienced a pulmonary embolus, deep venous thrombosis or other clinically significant thromboembolic event within 6 months of enrollment are eligible if they are clinically stable on anticoagulation therapy
* Current active infection, including known human immunodeficiency virus (HIV) positivity; for HIV patients on highly active antiretroviral therapy (HAART), the pharmacokinetics of the investigation agent may be seriously affected; when appropriate, 17-AAG will be studied in patients with HIV on HAART
* Pregnancy or breastfeeding; because of the unknown effects on the developing fetus/newborn, patients who are pregnant or become pregnant should be excluded from protocol study; exclusion of breast feeding women would also be appropriate as it is not known whether 17-AAG may be excreted in breast milk and what effect this may have on a developing newborn; female patients must agree to use effective contraception during the study period, be surgically sterile, or be post-menopausal; in addition, male patients will be required to use effective contraception during the study period or be surgically sterile; the definition of effective contraception will be based on the judgment of the investigator
* Serious allergy to eggs (i.e. hypotension, dyspnea, anaphylaxis, edema)
* Treatment with any agents that interact with cytochrome P450 3A should be avoided and used with caution, if necessary; when possible, patients should be switched to alternative medications; patients requiring anticoagulation should not be treated with Coumadin and should be switched to a low molecular weight heparin injection; patients receiving treatment with a low molecular weight heparin will require episodic monitoring with the anti-factor Xa heparin assay
* Previous (within 5 years of enrollment) or current malignancies at other sites, except adequately treated basal cell or squamous cell skin cancers and carcinoma in situ of the cervix
* Other severe acute or chronic medical or psychiatric conditions or laboratory abnormality that may increase the risk associated with study participation or study drug administration or may interfere with interpretation of study results and, in the judgment of the investigator, would make the patient inappropriate for study entry
* The use of concomitant medications that prolong or may prolong QTc are excluded
* Patients who have significant cardiac disease including heart failure that meets New York Heart Association (NYHA) class III and IV definitions, history of myocardial infarction within one year of study entry, uncontrolled dysrhythmias, or poorly controlled angina are excluded
* Patients who have a history of serious ventricular arrhythmia (VT or VF, >= 3 beats in a row), QTc >= 450 msec for men and 470 msec for women, or LVEF =< 40% by MUGA are excluded
* Patients with a prior history of cardiac or pulmonary toxicity after receiving anthracyclines such as doxorubicin, daunorubicin, mitoxantrone, bleomycin or BCNU
* Patients with greater or equal to grade 2 pulmonary or cardiac symptoms prior to study entry
* Patients with a history of prior radiation that potentially included the heart in the field (e.g., mantle)
* Patients with active ischemic heart disease within 12 months
* Patients with a history of uncontrolled dysrhythmias or requiring antiarrhythmic drugs
* Patients with congenital long QT syndrome; and patients with left bundle branch block
* Patients with symptomatic pulmonary disease requiring medication including the following: dyspnea, dyspnea on exertion, paroxysmal nocturnal dyspnea, oxygen requirement and significant pulmonary disease, including chronic obstructive/restrictive pulmonary disease
* Patients that meet the Medicare criteria for home oxygen
* Patients with a prior history of chest radiation

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2005-09; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elaina Gartner, Principal Investigator — Wayne State University
Locations (1):
- Barbara Ann Karmanos Cancer Institute, Detroit, Michigan, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Cancer center clinic.
Groups:
- Treatment (Tanespimycin): Patients receive tanespimycin IV over 1-6 hours on days 1, 4, 8, and 11. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.
  Laboratory biomarker analysis: Correlative studies (was not completed due to the small number of samples)
Period: Overall Study
Arm/Group | Treatment (Tanespimycin)
Started | 11
Completed | 11
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Tanespimycin)
Number analyzed (Participants) | 11
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 9
  >=65 years | 2
Gender [Count of Participants; unit: Participants]
  Female | 11
  Male | 0
Region of Enrollment [Number; unit: participants]
  United States | 11

OUTCOME MEASURES:

1. Primary Outcome: Response Rate (Complete Response (CR) +Partial Response (PR)
Description: Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR.
Time Frame: Up to 7 years
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Tanespimycin)
Number analyzed (Participants) | 7
Participants | 0

2. Primary Outcome: Progression Free Survival (PFS)
Description: PFS is defined as either progression or death, whichever occurs first. Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions.
Time Frame: Up to 7 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Treatment (Tanespimycin)
Number analyzed (Participants) | 11
months | 2 [1 to 11]

3. Primary Outcome: Her2/Neu Status
Description: Response rates will be estimated separately for her2/neu positive and her2/neu negative individuals along with 95% confidence intervals.
  PLEASE NOTE: IT WAS PROPOSED TO ANALYZE OUTCOME BY HER2 STATUS, NO DATA WAS COLLECTED OR EVALUATED.
Time Frame: Baseline
Population: No participants were evaluated for her2/neu status.
Arm/Group | Treatment (Tanespimycin)
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: 30 days after the last dose of treatment
Arm/Group | Treatment (Tanespimycin)
Serious Adverse Events (participants affected / at risk) | 6/11
Other Adverse Events (participants affected / at risk) | 9/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Tanespimycin) (N=11)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (1)
Hypotension (Vascular disorders) | 1 (1)
Fatigue (General disorders) | 1 (1)
Urinary Tract Infection (Infections and infestations) | 1 (1)
Lung Infection (Infections and infestations) | 1 (1)
Aspartate Aminotransferase Increased (Investigations) | 1 (1)
Alkaline Phosphatase Increased (Investigations) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 1 (1)
Anaphylaxis (Immune system disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Voice Alteration (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 1 (1)
Pleural Infection (Infections and infestations) | 1 (1)
Respiratory, Thoracic, and Mediastinal Disorders - Other, specify (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Alkaline Phosphatase Increased (Investigations) | 2 (2)
Blood Bilirubin Increased (Investigations) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Tanespimycin) (N=11)
Anemia (Blood and lymphatic system disorders) | 7 (11)
Anorexia (Metabolism and nutrition disorders) | 4 (6)
Sinus Tachycardia (Cardiac disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
Edema Limbs (General disorders) | 1 (1)
Lymphocyte Count Decreased (Investigations) | 3 (3)
Blood Bilirubin Increased (Investigations) | 2 (2)
Alanine Aminotransferase Increased (Investigations) | 3 (4)
Aspartate Aminotransferase (Investigations) | 5 (7)
Hyperglycemia (Metabolism and nutrition disorders) | 4 (7)
White Blood Cell Decreased (Investigations) | 2 (3)
Ventricular Arrhythmia (Cardiac disorders) | 1 (1)
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 1 (1)
Headache (Nervous system disorders) | 2 (2)
Diarrhea (Gastrointestinal disorders) | 3 (5)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Alkaline Phosphatase Increased (Investigations) | 3 (5)
Constipation (Gastrointestinal disorders) | 2 (2)
Confusion (Psychiatric disorders) | 1 (1)
Infections and Infestations - Other (Infections and infestations) | 1 (2)
Fatigue (General disorders) | 3 (4)
Nausea (Gastrointestinal disorders) | 3 (4)
Hepatobiliary Disorders - Other (Hepatobiliary disorders) | 1 (2)
Generalized Muscle Weakness (Musculoskeletal and connective tissue disorders) | 1 (1)
Hypermagnesemia (Metabolism and nutrition disorders) | 2 (4)
Hypocalcemia (Metabolism and nutrition disorders) | 2 (5)
Blurred Vision (Eye disorders) | 1 (2)
Bone Pain (Musculoskeletal and connective tissue disorders) | 1 (3)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (3)
Hypercalcemia (Metabolism and nutrition disorders) | 2 (3)
Body Odor (Skin and subcutaneous tissue disorders) | 1 (1)
Abdominal Pain (Gastrointestinal disorders) | 1 (1)
Urinary Tract Pain (Renal and urinary disorders) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1)
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 (2)
Hypokalemia (Metabolism and nutrition disorders) | 1 (1)
Peripheral Sensory Neuropathy (Nervous system disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
Because of the frequency of toxicities experienced by the pts & lack of response, study closed to accrual before all 17 planned pts were enrolled. It was proposed to analyze outcome by HER2 status,but no HER2 data was collected.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less